CLINICAL TRIAL: NCT01371656
Title: A Randomized Trial of Levofloxacin to Prevent Bacteremia in Children Being Treated for Acute Leukemia (AL) or Undergoing Hematopoietic Stem Cell Transplantation (HSCT)
Brief Title: Levofloxacin in Preventing Infection in Young Patients With Acute Leukemia Receiving Chemotherapy or Undergoing Stem Cell Transplantation
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: ACCL0934; NCI-2011-02636 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000695661 (Other: ClinicalTrials.gov); ACCL0934 (Other: Children's Oncology Group); COG-ACCL0934 (Other: DCP); ACCL0934 (Other: CTEP); U10CA095861 (NIH)
Record Dates: First submitted 2011-06-04; First posted 2011-06-13 (Estimated); Results first posted 2018-06-26 (Actual); Last update posted 2020-12-07 (Actual); Status verified 2018-06

CONDITIONS: Acute Leukemias of Ambiguous Lineage; Bacterial Infection; Diarrhea; Fungal Infection; Musculoskeletal Complications; Neutropenia; Recurrent Childhood Acute Lymphoblastic Leukemia; Recurrent Childhood Acute Myeloid Leukemia; Secondary Acute Myeloid Leukemia; Untreated Childhood Acute Myeloid Leukemia and Other Myeloid Malignancies
MeSH Terms: conditions — Leukemia, Biphenotypic, Acute; Bacterial Infections; Diarrhea; Mycoses; Neutropenia; Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Levofloxacin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (levofloxacin) (Experimental): Patients receive levofloxacin PO or IV over 60-90 minutes once or twice daily beginning on day 3 during 2 consecutive courses of chemotherapy or beginning on day -2 during HSCT and continuing until blood counts recover.
  Interventions: Drug: levofloxacin
- Arm II (standard of care) (No Intervention): Patients receive established standard of care and receive chemotherapy or HSCT as patients in Arm I.

INTERVENTIONS:
Drug: levofloxacin — Given PO or IV
  Other Names: Levaquin; Quixin
  Arms: Arm I (levofloxacin)

SUMMARY:
This randomized phase III trial studies how well levofloxacin works in preventing infection in young patients with acute leukemia receiving chemotherapy or undergoing stem cell transplant. Giving antibiotics may be effective in preventing or controlling early infection in patients receiving chemotherapy or undergoing stem cell transplant for acute leukemia. It is not yet known whether levofloxacin is effective in preventing infection.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine whether levofloxacin given prophylactically during periods of neutropenia to patients being treated with chemotherapy for acute leukemia (AL) or undergoing hematopoietic stem cell transplantation (HSCT) will decrease the incidence of bacteremia.

SECONDARY OBJECTIVES:

I. To determine the effect of prophylactic levofloxacin on resistance patterns of bacterial isolates from all sterile site cultures, and the evolution of antimicrobial resistance from peri-rectal swab isolates of Enterobacteriaceae, Escherichia coli, Klebsiella pneumoniae, Pseudomonas aeruginosa, and Streptococcus mitis.

II. To determine the effect of levofloxacin prophylaxis on total number of days of antibiotic administration (prophylactic, empiric, and treatment) in children undergoing therapy for AL or HSCT.

III. To determine whether levofloxacin prophylaxis reduces the incidence of fever with neutropenia, severe infection, and death from bacterial infection.

IV. To assess the safety of levofloxacin prophylaxis, with specific attention to musculoskeletal disorders including tendinopathy and tendon rupture.

V. To assess the impact of prophylactic levofloxacin on the incidence of Clostridium difficile-associated diarrhea (CDAD), and the incidence of microbiologically documented invasive fungal infections (IFI).

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

ARM I: Patients receive levofloxacin orally (PO) or intravenously (IV) over 60-90 minutes once daily (QD) or twice daily (BID) beginning on day 3 during 2 consecutive courses of chemotherapy or beginning on day -2 during HSCT and continuing until blood counts recover.

ARM II: Patients receive established standard of care and receive chemotherapy or HSCT as patients in Arm I.

After completion of study therapy, patients are followed up for 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Patient must fit 1 of the following 2 categories:

  * Chemotherapy patients

    * Planned to receive at least 2 consecutive cycles (not required to be the first 2 cycles) of intensive chemotherapy for either:

      * De novo, relapsed or secondary acute myeloid leukemia (AML), or acute leukemia of ambiguous lineage treated with standard AML therapy
      * Relapsed acute lymphoblastic leukemia (ALL)
      * For the purposes of this study, "intensive chemotherapy" is defined as regimens that are predicted by the local investigator to cause neutropenia for > 7 days; examples include, but are not limited to, treatment with "4-drug induction" (anthracycline, vincristine, asparaginase, and steroid), high dose cytarabine, anthracycline/cytarabine, ifosfamide/etoposide, and clofarabine-containing regimens
  * Stem cell transplantation patients

    * Planned to receive at least 1 myeloablative autologous or allogeneic HSCT
    * For the purposes of this study, myeloablative autologous and allogeneic HSCT are those in which the conditioning regimen is predicted by the local Investigator to cause neutropenia for > 7 days
* Creatinine clearance or radioisotope glomerular filtration rate (GFR) > 70 mL/min/1.73 m^2 OR serum creatinine based on age/gender as follows:

  * 0.5 mg/dL (6 months to < 1 year of age)
  * 0.6 mg/dL (1 to < 2 years of age)
  * 0.8 mg/dL (2 to < 6 years of age)
  * 1.0 mg/dL (6 to < 10 years of age)
  * 1.2 mg/dL (10 to < 13 years of age)
  * 1.5 mg/dL (male)/1.4 mg/dL (female) (13 to < 16 years of age)
  * 1.7 mg/dL (male)/1.4 mg/dL (female) (>= 16 years of age)
* Patients must have a performance status corresponding to Eastern Cooperative Oncology Group (ECOG) scores of 0, 1, or 2; use Karnofsky for patients > 16 years of age and Lansky for patients =< 16 years of age
* All patients and/or their parents or legal guardians must sign a written informed consent
* All institutional, Food and Drug Administration (FDA), and National Cancer Institute (NCI) requirements for human studies must be met

Exclusion Criteria:

* Patients previously enrolled on the trial are not eligible; therefore, patients with AL who were on study during intensive chemotherapy are not eligible to be enrolled during the HSCT
* Patients with an allergy to quinolones
* Patients with chronic active arthritis
* Patients with a known pathologic prolongation of the corrected QT (QTc)
* Females who are pregnant or breast feeding
* Patients being treated with antibacterial agents, other than any of the following:

  * Cotrimoxazole or other agents including dapsone, atovaquone, and pentamidine administered for Pneumocystitis jiroveci (PCP) prophylaxis
  * Topical antibiotics
  * Central venous catheter antibiotic lock therapy
  * Note: prophylactic antifungal therapy is NOT an exclusion criterion
* Patients currently enrolled on the ACCL1034 study are not eligible until they have completed the 90 day observation period of that study

Ages: 6 Months to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 624 (Actual)
Dates: Start 2011-09 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Alexander, MD, Principal Investigator — Children's Oncology Group
Locations (84):
- United States (78):
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - Southern California Permanente Medical Group, Downey, California
  - City of Hope Medical Center, Duarte, California
  - Loma Linda University Medical Center, Loma Linda, California
  - Miller Children's Hospital, Long Beach, California
  - Children's Hospital Los Angeles, Los Angeles, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Rady Children's Hospital - San Diego, San Diego, California
  - University of California San Francisco Medical Center-Parnassus, San Francisco, California
  - Connecticut Children's Medical Center, Hartford, Connecticut
  - Alfred I duPont Hospital for Children, Wilmington, Delaware
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Lombardi Comprehensive Cancer Center at Georgetown University, Washington D.C., District of Columbia
  - Golisano Children's Hospital of Southwest Florida, Fort Myers, Florida
  - Nemours Children's Clinic - Jacksonville, Jacksonville, Florida
  - Nemours Children's Hospital, Orlando, Florida
  - Nemours Children's Clinic - Pensacola, Pensacola, Florida
  - All Children's Hospital, St. Petersburg, Florida
  - Saint Mary's Hospital, West Palm Beach, Florida
  - Children's Healthcare of Atlanta - Egleston, Atlanta, Georgia
  - Georgia Regents University, Augusta, Georgia
  - University of Illinois, Chicago, Illinois
  - Advocate Children's Hospital-Oak Lawn, Oak Lawn, Illinois
  - Riley Hospital for Children, Indianapolis, Indiana
  - Saint Vincent Hospital and Health Services, Indianapolis, Indiana
  - Blank Children's Hospital, Des Moines, Iowa
  - University of Kentucky, Lexington, Kentucky
  - Kosair Children's Hospital, Louisville, Kentucky
  - Tulane University Health Sciences Center, New Orleans, Louisiana
  - Children's Hospital-Main Campus, New Orleans, Louisiana
  - Ochsner Medical Center, New Orleans, Louisiana
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - Floating Hospital for Children at Tufts Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - C S Mott Children's Hospital, Ann Arbor, Michigan
  - Helen DeVos Children's Hospital at Spectrum Health, Grand Rapids, Michigan
  - Michigan State University - Breslin Cancer Center, Lansing, Michigan
  - Children's Hospitals and Clinics of Minnesota - Minneapolis, Minneapolis, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Saint John's Mercy Medical Center, St Louis, Missouri
  - Children's Hospital and Medical Center of Omaha, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Nevada Cancer Research Foundation CCOP, Las Vegas, Nevada
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Saint Peter's University Hospital, New Brunswick, New Jersey
  - UMDNJ - Robert Wood Johnson University Hospital, New Brunswick, New Jersey
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Roswell Park Cancer Institute, Buffalo, New York
  - New York University Langone Medical Center, New York, New York
  - Columbia University Medical Center, New York, New York
  - University of Rochester, Rochester, New York
  - Montefiore Medical Center, The Bronx, New York
  - Ny Cancer%, Valhalla, New York
  - Mission Hospital-Memorial Campus, Asheville, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Children's Hospital Medical Center of Akron, Akron, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - The Children's Medical Center of Dayton, Dayton, Ohio
  - The Toledo Hospital/Toledo Children's Hospital, Toledo, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Lehigh Valley Hospital - Muhlenberg, Bethlehem, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - Palmetto Health Richland, Columbia, South Carolina
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - Driscoll Children's Hospital, Corpus Christi, Texas
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Brooke Army Medical Center, Fort Sam Houston, Texas
  - Cook Children's Medical Center, Fort Worth, Texas
  - Baylor College of Medicine, Houston, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Methodist Children's Hospital of South Texas, San Antonio, Texas
  - Childrens Hospital-King's Daughters, Norfolk, Virginia
  - Providence Sacred Heart Medical Center and Children's Hospital, Spokane, Washington
  - Madigan Army Medical Center, Tacoma, Washington
  - Marshfield Clinic, Marshfield, Wisconsin
- Canada (6):
  - CancerCare Manitoba, Winnipeg, Manitoba
  - Janeway Child Health Centre, St. John's, Newfoundland and Labrador
  - McMaster Children's Hospital at Hamilton Health Sciences, Hamilton, Ontario
  - Cancer Centre of Southeastern Ontario at Kingston General Hospital, Kingston, Ontario
  - Hospital for Sick Children, Toronto, Ontario
  - The Montreal Children's Hospital of the MUHC, Montreal, Quebec

REFERENCES:
- See also: Data Available: Select individual patient-level data from this trial can be requested from the NCTN/NCORP Data Archive — https://nctn-data-archive.nci.nih.gov/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm I (Levofloxacin) | Arm II (Standard of Care)
Started | 314 | 310
Completed | 250 | 296
Not Completed | 64 | 14
Not completed — Death | 7 | 4
Not completed — Physician Decision | 46 | 7
Not completed — Withdrawal by Subject | 7 | 0
Not completed — Ineligible | 4 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (Levofloxacin) | Arm II (Standard of Care) | Total
Number analyzed (Participants) | 314 | 310 | 624
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 275 | 284 | 559
  Between 18 and 65 years | 39 | 26 | 65
  >=65 years | 0 | 0 | 0
Age, Continuous [Median (Standard Deviation); unit: Years] | 9.44 (6.18) | 9.18 (5.89) | 9.31 (6.03)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 120 | 127 | 247
  Male | 194 | 183 | 377
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 89 | 56 | 145
  Not Hispanic or Latino | 208 | 246 | 454
  Unknown or Not Reported | 17 | 8 | 25
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 22 | 17 | 39
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 35 | 45 | 80
  White | 217 | 216 | 433
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 40 | 32 | 72
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 287 | 272 | 559
  Canada | 26 | 36 | 62
  India | 1 | 0 | 1
  Mexico | 0 | 1 | 1
  Ireland | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Comparison of the Percentage of Patients Having Bacteremia Incidence Between Levofloxacin vs. No Prophylaxis Arms
Description: A bacteremia incidence is defined as an occurrence of at least 1 episode of true (centrally reviewed) bacteremia among Acute Leukemia (AL) and Hematopoietic stem cell transplantation (HSCT) patients.
Time Frame: Up to 60 days after enrollment or receiving levofloxacin
Population: All evaluable, and centrally reviewed AL and HSCT patients are reported. Ineligible patients and patients who withdrew of consent prior to treatment were excluded.
Measure: Number; unit: Percentage of patients
Arm/Group | Arm I (Levofloxacin) | Arm II (Standard of Care)
Number analyzed (Participants) | 306 | 307
Percentage of patients
  Evaluable AL patients: number analyzed (Participants) | 96 | 99
  Evaluable AL patients | 21.9 | 43.4
  Evaluable HSCT patients: number analyzed (Participants) | 210 | 208
  Evaluable HSCT patients | 11 | 17.3

2. Secondary Outcome: Comparison of the Percentage of Patients Having Antibiotic Exposures Between Arms
Description: Exposure to antibiotics was considered during the infection observation period(s) was defined a priori as follows: Gram positive agents = vancomycin, linezolid, daptomycin or quinupristin/dalfopristin; Aminoglycosides = amikacin, gentamicin or tobramycin; Third or fourth generation cephalosporins = cefepime, ceftazidime, ceftriaxone or cefotaxime; Empiric antibiotics for fever and neutropenia = imipenem, meropenem, cefepime, ceftazidime or piperacillin/tazobactam
Time Frame: Up to 60 days after enrollment or receiving levofloxacin
Population: as for outcome 1
Measure: Number; unit: Percentage of patients
Arm/Group | Arm I (Levofloxacin) | Arm II (Standard of Care)
Number analyzed (Participants) | 306 | 307
Percentage of patients
  Gram positive agents | 58.8 | 65.8
  Aminoglycosides | 22.9 | 35.5
  Third or fourth generation cephalosporins | 46.1 | 59.9
  Empiric antibiotics for fever and neutropenia | 68.6 | 85.7

3. Secondary Outcome: Comparison of the Percentage of Patients Having Incidence of Fever and Febrile Neutropenia Between Arms
Description: Fever and febrile neutropenia defined as Absolute Neutrophil Count (ANC) < 1000/mm3 with a single temperature of >38.3 degrees C (101 degrees F) or a sustained temperature of >= 38 degrees C (100.4 degrees F) for more than one hour.
Time Frame: Up to 60 days after enrollment or receiving levofloxacin
Population: as for outcome 1
Measure: Number; unit: Percentage of patients
Arm/Group | Arm I (Levofloxacin) | Arm II (Standard of Care)
Number analyzed (Participants) | 306 | 307
Percentage of patients | 71.2 | 82.1

4. Secondary Outcome: Comparison of the Percentage of Patients Having Severe Infection Between Arms
Description: Severe infection defined as any grade 4 or 5 CTCAE catheter-related infection, enterocolitis, lung infection, sepsis, small intestine infection and other infections or infestations
Time Frame: Up to 60 days after enrollment or receiving levofloxacin
Population: as for outcome 1
Measure: Number; unit: Percentage of patients
Arm/Group | Arm I (Levofloxacin) | Arm II (Standard of Care)
Number analyzed (Participants) | 306 | 307
Percentage of patients | 3.6 | 5.9

5. Secondary Outcome: Comparison of the Percentage of Patients That Died Due to Bacterial Infection Between Arms
Time Frame: Up to 60 days after enrollment or receiving levofloxacin
Population: Evaluable patients combined from both AL and HSCT cohorts were reported. Ineligible and withdrew of Consent prior to Tx were excluded.
Measure: Number; unit: Percentage of patients
Arm/Group | Arm I (Levofloxacin) | Arm II (Standard of Care)
Number analyzed (Participants) | 306 | 307
Percentage of patients | 0 | 0

6. Secondary Outcome: Comparison of the Percentage of Patients Having Incidence of Musculoskeletal Adverse Events Including Tendinopathy (Tendonitis and Tendon Rupture) Between Arms
Description: Musculoskeletal conditions included at least one occurrence of arthralgia, arthritis, gait abnormality or tendinopathy.
Time Frame: Enrollment, 2 months and 12 months post infection observation period
Population: Evaluable patients who submitted musculoskeletal Case Record Form (CRF) combined from both Acute Leukemia (AL) and Hematopoietic stem cell transplantation (HSCT) cohorts at enrollment. Ineligible and withdrew of Consent prior to treatment were excluded.
Measure: Number; unit: Percentage of patients
Arm/Group | Arm I (Levofloxacin) | Arm II (Standard of Care)
Number analyzed (Participants) | 303 | 300
Percentage of patients
  Evaluable AL and HSCT Patients at Baseline | 5.9 | 10
  Evaluable AL and HSCT Patients at 2 Months: number analyzed (Participants) | 201 | 240
  Evaluable AL and HSCT Patients at 2 Months | 11.4 | 16.3
  Evaluable AL and HSCT Patients at 12 Months: number analyzed (Participants) | 129 | 146
  Evaluable AL and HSCT Patients at 12 Months | 10.1 | 14.4

7. Secondary Outcome: Comparison of the Percentage of Patients Having Incidence of CDAD Between Arms
Description: Clostridium Difficile Associated Disease (CDAD) is defined as a positive C. difficile toxin assay result and diarrhea, CTCAE version 4, grade 2 and higher.
Time Frame: Up to 60 days after enrollment or receiving levofloxacin
Population: as for outcome 1
Measure: Number; unit: Percentage of patients
Arm/Group | Arm I (Levofloxacin) | Arm II (Standard of Care)
Number analyzed (Participants) | 306 | 307
Percentage of patients | 2.3 | 5.2

ADVERSE EVENTS:
Time Frame: Up to 60 days after enrollment or receiving of levofloxacin
Description: Routine reporting includes all toxicities reported via AdEERs and all grade 4 & higher non-hematologic Adverse Events
Arm/Group | Arm I (Levofloxacin) | Arm II (Standard of Care)
All-Cause Mortality (participants affected / at risk) | 69/306 | 67/307
Serious Adverse Events (participants affected / at risk) | 4/306 | 3/307
Other Adverse Events (participants affected / at risk) | 36/306 | 37/307
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I (Levofloxacin) (N=306) | Arm II (Standard of Care) (N=307)
Acute kidney injury (Renal and urinary disorders) | 1 | 0
Capillary leak syndrome (Vascular disorders) | 1 | 0
Death NOS (General disorders) | 1 | 1
Heart failure (Cardiac disorders) | 0 | 1
Infections and infestations - Other, specify (Infections and infestations) | 2 | 0
Lung infection (Infections and infestations) | 0 | 1
Multi-organ failure (General disorders) | 3 | 0
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Sepsis (Infections and infestations) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I (Levofloxacin) (N=306) | Arm II (Standard of Care) (N=307)
Acidosis (Metabolism and nutrition disorders) | 0 | 2
Acute kidney injury (Renal and urinary disorders) | 1 | 1
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Alanine aminotransferase increased (Investigations) | 3 | 4
Alkalosis (Metabolism and nutrition disorders) | 0 | 1
Anaphylaxis (Immune system disorders) | 1 | 0
Aspartate aminotransferase increased (Investigations) | 2 | 2
Asystole (Cardiac disorders) | 0 | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Blood bilirubin increased (Investigations) | 3 | 2
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Capillary leak syndrome (Vascular disorders) | 1 | 0
Cardiac arrest (Cardiac disorders) | 0 | 2
Catheter related infection (Infections and infestations) | 0 | 1
Depressed level of consciousness (Nervous system disorders) | 0 | 1
Diarrhea (Gastrointestinal disorders) | 1 | 0
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Encephalopathy (Nervous system disorders) | 0 | 1
Enterocolitis infectious (Infections and infestations) | 0 | 1
Fibrinogen decreased (Investigations) | 1 | 0
GGT increased (Investigations) | 2 | 3
Hepatic failure (Hepatobiliary disorders) | 0 | 1
Hepatobiliary disorders - Other, specify (Hepatobiliary disorders) | 2 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 4 | 2
Hyperkalemia (Metabolism and nutrition disorders) | 0 | 1
Hypernatremia (Metabolism and nutrition disorders) | 0 | 1
Hypertriglyceridemia (Metabolism and nutrition disorders) | 2 | 0
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 | 1
Hypocalcemia (Metabolism and nutrition disorders) | 1 | 3
Hypokalemia (Metabolism and nutrition disorders) | 3 | 5
Hypomagnesemia (Metabolism and nutrition disorders) | 0 | 1
Hyponatremia (Metabolism and nutrition disorders) | 1 | 2
Hypotension (Vascular disorders) | 3 | 4
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Ileal hemorrhage (Gastrointestinal disorders) | 0 | 1
Infections and infestations - Other, specify (Infections and infestations) | 1 | 4
Intracranial hemorrhage (Nervous system disorders) | 0 | 1
Left ventricular systolic dysfunction (Cardiac disorders) | 0 | 1
Lung infection (Infections and infestations) | 0 | 1
Mucositis oral (Gastrointestinal disorders) | 2 | 4
Multi-organ failure (General disorders) | 0 | 1
Nervous system disorders - Other, specify (Nervous system disorders) | 0 | 1
Neutrophil count decreased (Investigations) | 0 | 1
Pericardial effusion (Cardiac disorders) | 1 | 0
Platelet count decreased (Investigations) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Portal hypertension (Hepatobiliary disorders) | 1 | 0
Portal vein thrombosis (Hepatobiliary disorders) | 0 | 1
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 1 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 5
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Reversible posterior leukoencephalopathy syndrome (Nervous system disorders) | 1 | 0
Seizure (Nervous system disorders) | 0 | 1
Sepsis (Infections and infestations) | 8 | 11
Sinus bradycardia (Cardiac disorders) | 0 | 1
Small intestine infection (Infections and infestations) | 0 | 1
Stridor (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Ventricular fibrillation (Cardiac disorders) | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Must obtain prior Sponsor approval.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-01-27): https://cdn.clinicaltrials.gov/large-docs/56/NCT01371656/Prot_SAP_000.pdf